CLINICAL TRIAL: NCT05833971
Title: A Single-arm, Multicenter, Exploratory Study of Cadonilimab in Combination With Chemotherapy for Locally Advaced Esophageal Squamous Cell Carcinoma
Brief Title: Cadonilimab in Combination With Chemotherapy for Locally Advaced Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jun Liu, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cadonilimab-Neoadjuvant
Record Dates: First submitted 2023-02-25; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: cadonilimab (AK104) + chemotherapy (Experimental): Drug: Cadonilimab+ chemotherapy，10mg/kg IV every 3 weeks (Q3W)，Other Name: AK104； Cisplatin，60-75mg/m2 IV every 3 weeks (Q3W)，Other Name: DDP；Albumin Paclitaxel，260mg/m2 IV every 3 weeks D1, 8(Q3W)，Other Name: Nab-PTX
  Interventions: Drug: cadonilimab+chemotherapy

INTERVENTIONS:
Drug: cadonilimab+chemotherapy — cadonilimab plus cisplatin and Nab-PTX, Q3W
  Other Names: AK104

SUMMARY:
This is a single-arm, multicenter, exploratory study to evaluate the efficacy and safety of AK104 in combination with cisplatin and paclitaxel in the treatment of resectable locally advanced esophageal squamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years, both men and women
* Pathologically confirmed esophageal squamous cell carcinoma，and the clinic staging is cT2N1-3M0 or cT3N0-3M0 or cT4N0-3M0, TNM staging is II-IVA
* Non-cervical esophageal carcinoma
* Patients who have never received systemic antitumor therapy and who have measurable lesions that meet RECIST 1.1 criteria
* ECOG score 0-1
* Life expectancy ≥12 months
* Patients with normal function organs, no serious abnormalities of blood, heart, lung, liver, kidney function, and immunodeficiency disease
* For female subjects of childbearing age, they should have a negative urine or serum pregnancy test within 7 days before receiving the first study drug administration. Male and female patients need to use high-efficiency contraception during treatment until at least 8 weeks after stop the treatment
* Sign the informed consent form before any trial-related procedures are implemented

Exclusion Criteria:

* -Other malignancies diagnosed within 5 years prior to the first administration of the study drug, except effectively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or effectively resected in situ cervical and/or breast cancer
* ulcerative esophageal squamous cell carcinoma
* Esophageal or tracheal fistula
* History of allergy to study drug components
* History of immune disease
* Patients with any serious or uncontrolled systemic disease
* The presence of any adverse event (CTCAE>grade 1) caused by prior therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) | 1 month after resection
  Analysis of prognosis efficacy of patients: pathologic complete response (pCR)

SECONDARY OUTCOMES:
Radical resection (R0) | 1 month after resection
Overall survival(OS) | up to 2 years
Objective response rate(ORR) | After the start of drugs and before resection
Disease control rate(DCR) | After the start of drugs and before resection
Disease-free survival(DFS) | After resection and up to 2 years

IPD SHARING:
Plan to Share IPD: No